CLINICAL TRIAL: NCT07338903
Title: Move to Improve: Investigating the Feasibility of Embedding Physical Activity Into Routine Breast Cancer Care in Indonesia
Brief Title: Feasibility and Effects of Home-based Physical Activity Intervention in Patients With Breast Cancer in Indonesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Collaborators: University of Leeds (Other); Durham University (Other)
Responsible Party: Principal Investigator, Susanna Hilda Hutajulu, Susanna Hilda Hutajulu, MD, PhD, Gadjah Mada University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 3550/UN1.P.III/DitLit/PT.01.05
Record Dates: First submitted 2026-01-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Breast Neoplasms; Physical Fitness
Keywords: Breast neoplasms; Physical activity; Exercise; Walking; Resistance exercise; Physical fitness; Fatigue; Quality of life
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical activity intervention (Experimental)
  Interventions: Behavioral: 12weeks of home-based aerobic (pedometer-driven walking) and resistance training using therapeutic bands

INTERVENTIONS:
Behavioral: 12weeks of home-based aerobic (pedometer-driven walking) and resistance training using therapeutic bands — 1. Home-based aerobic training: The aerobic exercise consisted of a walking program based on the number of steps per day, which was recorded using a pedometer (Yamax Digiwalker SW-200, Tokyo, Japan). The target of the aerobic exercise was individually tailored by adding 3000 accumulated steps above their baseline value on 5 days of the week.
  2. Home-based resistance training: The resistance training was conducted using a set of resistance bands (Happy Fit®, Jakarta, Indonesia). This training consisted of two sets of biceps curl, triceps extension, chest press, shoulder flexion, shoulder press, lateral extension, seated row, and upright row, with 8-10 repetitions. Patients were instructed to perform each exercise with an average total duration of 10 minutes on 2 days a week at home. The exercises were individually tailored based on participants' strength and range of movement using a set of three color-coded bands representing low, moderate, and high levels of resistance.

SUMMARY:
The goal of this clinical trial is to learn the impact and implementation of home-based aerobic and resistance training for patients with breast cancer in Indonesia. The main questions it aims to answer are:

* Does the home-based aerobic and resistance training improve physical fitness, fatigue, and quality of life of patients with breast cancer?
* Are the benefits of aerobic and resistance training mediated by inflammatory level changes?
* What are the barriers and facilitators in implementing the home-based aerobic and resistance training?
* Is the home-based aerobic and resistance training feasible to be implemented in Indonesia's setting?

To answer those questions, participants will:

* Conduct home-based aerobic and resistance training with supervision.
* Visit the hospital once every 4 weeks for their routine visits.
* Undergo physical fitness test before and after 12 weeks using treadmill test, as well as interviews to assess fatigue, quality of life, and intervention acceptability.
* Keep a diary to record the aerobic and resistance training at home.
* Undergo routine monitoring by phone every week with the research team.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage I-III hormone-receptor positive breast cancer
* Eastern Cooperative Oncology Group (ECOG) score ≤1
* Had completed primary treatment (e.g., surgery, chemotherapy, and radiotherapy), except for hormonal treatment
* Within 5 years of diagnosis
* Able to perform moderate-intensity physical activity as determined by their oncologist and care team
* Able to read and write in Indonesian
* Willing to provide written informed consent.

Exclusion Criteria:

* Had an ejection fraction of <50%
* Evidence of cardiac disease, severe musculoskeletal problems, or other contraindications for exercise.

Ages: 17 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Physical fitness | Baseline and post-intervention (12 weeks)
  Physical fitness was measured using a submaximal treadmill test with the modified Bruce protocol. Treadmill speed and inclination were automatically increased every 3 min (test stage). The test was terminated when participants reached volitional fatigue. Physical fitness was classified as low, fair, average, and good, based on patients' age, treadmill test duration, and predicted VO2peak.
Fatigue | Baseline and post-intervention (12 weeks)
  Fatigue was assessed using the Indonesian version of Fatigue Severity Scale (FSS). A higher score on the FSS indicated a more severe level of fatigue. The FSS was also classified as no-to-mild fatigue (FSS <4.0) and severe fatigue (≥4.0).
Health-related quality of life | Baseline and post-intervention (12 weeks)
  Health-related quality of life was assessed using the Indonesian version of the EORTC Quality of Life Questionnaire (QLQ-C30). The EORTC QLQ-C30 consists of global health status, functional scales, and symptom scales. A higher score indicates better health for global health status and functional scales, but represents a higher level of burden for symptom scales.

SECONDARY OUTCOMES:
Inflammatory biomarkers | Baseline and post-intervention (12 weeks)
  Venous blood (5 ml) was collected at baseline and post-intervention to measure the levels of inflammatory biomarkers, including CRP, IL-6, and IL-10. The CRP levels were measured using an Enzyme-Linked Immunosorbent Assay (ELISA) assay (Calbiotech, CR120C), while IL-6 and IL-10 were measured using a Luminex assay (eBioscience, PPX-02-MXYMMK2).
Intervention acceptability | Post-intervention (12 weeks)
  Intervention acceptability was explored using semi-structured interviews using a research team-developed interview guide. All interviews were individual and face-to-face, took place in a private room, and were audiotaped.
Intervention barriers and facilitators | Post-intervention (12 weeks)
  Intervention barriers and facilitators were explored using semi-structured interviews using research team-developed interview guide. All interviews were individual and face-to-face, took place in a private room, and audiotaped.

OTHER OUTCOMES:
Intervention feasibility | During study period (baseline to 12 weeks)
  Intervention feasibility was determined by (a) recruitment (ratio of the number of participants recruited to the number of eligible participants approached), (b) retention (ratio of the number of participants who completed the 12-week program to the total number of participants enrolled in the study), (c) adherence (the ratio of the number of participants meeting at least 70% of prescribed activities calculated using steps per day, resistance exercise frequency, duration, and intensity to the total number of participants completing the 12-week program). The intervention was defined as feasible if those rates were above 75%.
Adverse events | During study period (baseline to 12 weeks)
  Adverse events (e.g., dyspnea, tachycardia, nausea, pain, and myalgia) that were reported by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Susanna H Hutajulu, MD, PhD, Principal Investigator — Faculty of Medicine, Public Health and Nursing, Universitas Gadjah Mada/Dr. Sardjito General Hospital; Shaunna Burke, PhD, Study Chair — Faculty of Biological Sciences, School of Biomedical Sciences, University of Leeds
Locations (1):
- Dr. Sardjito General Hospital, Sleman, Yogyakarta Special Region, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
The IPD that underlie results in the publication are accessible from the corresponding author upon reasonable request and subject to applicable data sharing agreements and approval processes.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Leite VF, Cecatto RB, Battistella LR, de Brito CMM. Establishing a Cancer Rehabilitation Service in a Middle-Income Country: an Experience from Brazil. Curr Phys Med Rehabil Rep. 2022;10(4):339-344. doi: 10.1007/s40141-022-00373-4. Epub 2022 Nov 28. PMID 36466557
- [Background] Batalik L, Winnige P, Dosbaba F, Vlazna D, Janikova A. Home-Based Aerobic and Resistance Exercise Interventions in Cancer Patients and Survivors: A Systematic Review. Cancers (Basel). 2021 Apr 15;13(8):1915. doi: 10.3390/cancers13081915. PMID 33921141
- [Background] de Jesus Leite MAF, Puga GM, Arantes FJ, Oliveira CJF, Cunha LM, Bortolini MJS, Penha-Silva N. Effects of combined and resistance training on the inflammatory profile in breast cancer survivors: A systematic review. Complement Ther Med. 2018 Feb;36:73-81. doi: 10.1016/j.ctim.2017.11.023. Epub 2017 Dec 1. PMID 29458936
- [Background] Lahart IM, Metsios GS, Nevill AM, Carmichael AR. Physical activity for women with breast cancer after adjuvant therapy. Cochrane Database Syst Rev. 2018 Jan 29;1(1):CD011292. doi: 10.1002/14651858.CD011292.pub2. PMID 29376559
- [Background] McNeely ML, Campbell KL, Rowe BH, Klassen TP, Mackey JR, Courneya KS. Effects of exercise on breast cancer patients and survivors: a systematic review and meta-analysis. CMAJ. 2006 Jul 4;175(1):34-41. doi: 10.1503/cmaj.051073. PMID 16818906